CLINICAL TRIAL: NCT02787889
Title: Effect of Dietary Protein Intake Distribution on Protein Metabolism and Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 139057
Record Dates: First submitted 2016-05-12; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uneven Protein Intake Pattern (Experimental): Subjects consumed either dietary protein intake at 1.1g protein/kg/day over 8 weeks.Each participant will consume 15%/2-%/65% of total protein in breakfast, lunch, and dinner, respectively)] on net protein synthesis over 8 weeks.
  Interventions: Other: Uneven Protein intake pattern
- Even Protein Intake Pattern (Experimental): Subjects consumed either dietary protein intake at 1.1g protein/kg/day over 8 weeks. Each participant will consume 33% of total protein consumed each meal
  Interventions: Other: Even Protein Intake Pattern

INTERVENTIONS:
Other: Uneven Protein intake pattern — Each participant will consume 15%/2-%/65% of total protein in breakfast, lunch, and dinner, respectively)] on net protein synthesis over 8 weeks.
  Arms: Uneven Protein Intake Pattern
Other: Even Protein Intake Pattern — Each participant will consume 33% of total protein consumed each meal
  Arms: Even Protein Intake Pattern

SUMMARY:
The investigators determined effects of 8-week dietary protein intake in mixed meals with uneven or even consumption pattern on the metabolic outcomes of whole-body net protein synthesis and muscle protein synthesis in older participants.

DETAILED DESCRIPTION:
The demonstrated benefits of increased protein intake on sarcopenia and many physiological functions is becoming increasingly evident. For this reason, there is growing importance to ensuring that Americans consume the recommended amount of protein, calculated to be 17-21% of caloric intake. As it relates to the prevention of sarcopenia, adequate protein consumption inherently assumes that sufficient protein is ingested to stimulate protein anabolism. Specifically, adequate essential amino acid precursors, and anabolic triggers such as leucine, must be present for protein anabolism to occur. Population data from the NHANES study suggests that American protein intake pattern is skewed towards the evening meal. The NHANES data also suggests that the average protein consumption of both men and women over the age of 50 yrs is approximately 1.1 g/kg/d. Thus, the prevalent consumption pattern ensures that many individuals consume adequate protein, or amino acid precursors sufficient to stimulate protein synthesis, only with the larger, or dinner meal. The investigators have demonstrated that frequent stimulation of protein synthesis with amino acids preserves strength and function. Others have demonstrated that adequate protein intake stimulates muscle protein synthesis and increases lean mass. Given these data, The investigators studied the effects of two different protein intake patterns on metabolic and functional outcomes in older individuals after 8 wks of dietary control. The mean protein intake for this group of 1.1 g/kg/d was consumed in two distinct meal patterns. Participants consumed high quality protein in the ratio of 15/20/65% of total protein intake for breakfast/lunch/dinner, respectively (Uneven protein intake pattern), or protein consumption was distributed equally among each meal (33% of total protein)(Even protein intake pattern). The investigators determined the longitudinal effects of this consumption pattern on the metabolic outcomes of whole-body net protein synthesis and muscle protein synthesis in older participants.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 50-70 years
* BMI between 24 and 30 kg/m2

Exclusion Criteria:

* Current diagnosis of diabetes
* History of malignancy in the 6 months prior to enrollment
* History of lactose intolerance or dairy allergy
* History of egg allergy or intolerance
* History of gastrointestinal bypass surgery.
* History of a chronic inflammatory condition or other chronic disease (Lupus, HIV/AIDS, etc)
* Subjects who do not or will not eat animal proteins
* Subjects who cannot refrain from consuming protein or amino acid supplements during their participation in this study
* Subjects who report regular resistance exercise (more than twice per week)
* Hemoglobin less than 9.5 mg/dL at the screening visit
* Platelets less than 150,000 at the screening visit
* Concomitant use of corticosteroids (ingestion, injection or transdermal)
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in net protein synthesis rate | Change from Baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arny A Ferrando, Ph.D., Principal Investigator — University of Arkansas

REFERENCES:
- [Derived] Kim IY, Schutzler S, Schrader AM, Spencer HJ, Azhar G, Wolfe RR, Ferrando AA. Protein intake distribution pattern does not affect anabolic response, lean body mass, muscle strength or function over 8 weeks in older adults: A randomized-controlled trial. Clin Nutr. 2018 Apr;37(2):488-493. doi: 10.1016/j.clnu.2017.02.020. Epub 2017 Mar 3. PMID 28318687